CLINICAL TRIAL: NCT05310032
Title: A Randomized, Open-label or Double-blind, Placebo Controlled, Single and Multiple Dosing, Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Food Effect After Oral Administration of HSG4112 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Food Effect of HSG4112 in High Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P1-04
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HSG4112 800 mg Single Dose (Experimental): Single oral dosing of HSG4112 800 mg
  Interventions: Drug: HSG4112
- HSG4112 1200 mg Single Dose (Experimental): Single oral dosing of HSG4112 1200 mg with a high-fat meal or fasting condition, with a washout period of 21 days in between each dosing
  Interventions: Drug: HSG4112
- HSG4112 800 mg Multiple Dose (Experimental): Multiple oral dosing of HSG4112 1200 mg for 14 days
  Interventions: Drug: HSG4112
- Placebo 800 mg Multiple Dose (Placebo Comparator): Multiple oral dosing of placebo 800 mg for 14 days
  Interventions: Drug: Placebo
- HSG4112 1200 mg Multiple Dose (Experimental): Multiple oral dosing of HSG4112 1200 mg for 14 days
  Interventions: Drug: HSG4112
- Placebo 1200mg Multiple Dose (Placebo Comparator): Multiple oral dosing of placebo 1200 mg for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSG4112 — Once-daily oral adminstration
  Other Names: 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: HSG4112 1200 mg Multiple Dose; HSG4112 1200 mg Single Dose; HSG4112 800 mg Multiple Dose; HSG4112 800 mg Single Dose
Drug: Placebo — Once-daily oral adminstration
  Arms: Placebo 1200mg Multiple Dose; Placebo 800 mg Multiple Dose

SUMMARY:
1. Study Objective

   i) To evaluate the safety, tolerability and pharmacokinetic/pharmacodynamic characteristics of HSG4112 after single and multiple oral administration of high doses in healthy subjects.

   ii) To evaluate the food effect on the pharmacokinetic characteristics of HSG4112 after a single oral administration of 1200 mg (6 tablets of HSG4112 200 mg) in healthy subjects.
2. Background

   The previous phase 1 clinical trials investigating HSG4112 included dosage only up to 720 mg of HSG4112 in both healthy and obese subjects. Since obese patients have various comorbidities, unexpected drug interactions may occur due to concomitant drugs. Securing a 2- to 5-fold safety margin is needed to tolerate this issue. Therefore, this study is designed to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics and food effects of high-dose HSG4112 in healthy subjects.
3. Study Design and Plan

<Part 1> This study is a randomized, open-label, single dosing, phase 1 clinical study. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. Each subject will be randomized to one of the two dose groups. 8 subjects will receive 800 mg of HSG4112 with a high-fat meal, and 12 subjects will be randomized to 2 different sequential groups. Each subject will receive a single dose of HSG4112 1200 mg via oral administration with a high-fat meal and in fasted condition, with a washout period of 21 days in between each dosing. When escalating the dose, the Investigator will review all of the available safety data from the preceding dose in a blinded manner to ensure if it is safe to escalate the dose. In order to evaluate safety and tolerability, assessments, such as vital signs, 12-lead ECG, laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed. Blood samples will be collected to evaluate the pharmacokinetic/pharmacodynamic characteristics of HSG4112.

<Part 2> This study is a randomized, double-blind, placebo-controlled, multiple dosing, phase 1 clinical study. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. Each subject will be randomized to one of the two dose groups (800 mg or 1200 mg of HSG4112). In each dose group, 6 subjects will be randomized to receive 800 mg of HSG4112, and 2 subjects will be randomized to receive placebo, both with a high-fat meal. The subjects will be studied in a double-blind manner and will receive the investigational product (i.e., HSG4112 or placebo) via once-daily oral administration for 14 days. When escalating the dose, the Investigator will review all of the available safety data from the preceding dose in a blinded manner to ensure if it is safe to escalate the dose. In order to evaluate safety and tolerability, assessments, such as vital signs, 12-lead ECG, laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed. Blood samples will be collected to evaluate the pharmacokinetic/pharmacodynamic characteristics of HSG4112.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before screening.
2. Adults between 19 and 50 years of age at screening.
3. Body mass index (BMI) between 18 and 24.9.

   * BMI (kg/m2) = Body weight (kg) / {Height (m)2}
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory test at screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.
5. For Part 2 (i.e., the multiple dose study), female subjects who have regular menstrual cycles(28±7 days) and who are not pregnant or lactating.

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, cardiovascular disease, or psychiatric disorder (e.g., mood disorder, obsessive-compulsive disorder).
2. History of stomach or intestinal disorders (e.g., Chrons disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the pharmacokinetic or pharmacodynamic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug compound (e.g., licorice-containing drugs, aspirin, antibiotics).
4. One or more of the following laboratory test results at screening:

   * ALT (SGPT) > 60 IU/L
   * Glucose (fasting) > 110 mg/dL or < 70 mg/dL
5. Systolic blood pressure of < 90 mmHg or > 150 mmHg, or diastolic blood pressure of < 60 mmHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for at least 3 minutes.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Use or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins within 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study involving the administration of an investigational drug, including any study investigating HSG4112, within 6 months prior to dosing (i.e., within 6 months of the last dose from the previous study).
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Smoker. However, participation is acceptable if the subject has quit smoking at least 90 days prior to dosing.
11. Alcohol consumption of > 21 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol during the study period, starting from 3 days prior to dosing.
12. Ingestion of grapefruit-containing foods or beverages 24 hours prior to dosing until discharge, or unable to abstain from ingesting such foods or beverages during the same period.
13. Unable to abstain from caffeine-containing foods or beverages (e.g., coffee, tea (e.g., black tea, green tea), soft drinks, coffee milk, energy drinks, sports drinks) during the admission period.
14. Unable or unwilling to use acceptable contraceptive methods for themselves or their spouse/partner during the entire study period and up to 28 days after the last dosing and subjects who satisfy at least one of the pregnancy-related criteria below:

    * females of childbearing potential who plan to use hormonal contraceptives or oral contraceptives during the study period
    * females of childbearing potential confirmed "positive" in a pregnancy test

      * "females of childbearing potential" refer to females who have experienced menarche and have not undergone a successful surgical sterilization procedure (i.e., hysterectomy, bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy) or is not menopause (i.e., 12 months without menstruation).

        * Acceptable contraceptive methods include:

          1. Use of an intrauterine device, which has been proven highly effective.
          2. Physical contraception for subject or spouse/partner used with chemical sterilization (e.g., spermicide).
          3. Surgical sterilization (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy).
15. Subjects who, in the opinion of the Investigator, should not participate in this study based on clinical laboratory test results or other reasons.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment by Maximum Plasma Concentration of HSG4112 | Hour 0 to 192
  Maximum Plasma Concentration of HSG4112 (Cmax)
Pharmacokinetic Assessment by Maximum Plasma Concentration of HSG4112 at Steady State | Hour 0 to 192
  Maximum Plasma Concentration of HSG4112 at Steady State (Cmax,ss)
Pharmacokinetic Assessment by Minimum Plasma Concentration of HSG4112 at Steady State | Hour 0 to 192
  Minimum Plasma Concentration of HSG4112 at Steady State (Cmin,ss)
Pharmacokinetic Assessment by Average Plasma Concentration of HSG4112 at Steady State | Hour 0 to 192
  Average Plasma Concentration of HSG4112 at Steady State (Cavg,ss)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity | Hour 0 to 192
  Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity (AUCinf)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity at Steady State | Hour 0 to 192
  Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity at Steady State (AUCinf,ss)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval | Hour 0 to 24
  Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval (AUCtau)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval at Steady State | Hour 0 to 24
  Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval at Steady State (AUCtau,ss)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point | Hour 0 to 192
  Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point (AUClast)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point at Steady State | Hour 0 to 192
  Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point at Steady State (AUClast,ss)
Pharmacokinetic Assessment by Half-Life of HSG4112 | Hour 0 to 192
  Half-life of HSG4112 (T1/2)
Pharmacokinetic Assessment by Half-Life of HSG4112 at Steady State | Hour 0 to 192
  Half-life of HSG4112 at Steady State (T1/2,ss)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HSG4112 | Hour 0 to 192
  Time to Maximum Observed Plasma of HSG4112 (Tmax)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HSG4112 at Steady State | Hour 0 to 192
  Time to Maximum Observed Plasma Concentration of HSG4112 at Steady State (Tmax,ss)
Pharmacokinetic Assessment by Oral Clearance of HSG4112 | Hour 0 to 192
  Oral Clearance of HSG4112 (CL/F)
Pharmacokinetic Assessment by Oral Clearance of HSG4112 at Steady State | Hour 0 to 192
  Oral Clearance of HSG4112 at Steady State (CLss/F)
Pharmacokinetic Assessment by Volume of Distribution of HSG4112 | Hour 0 to 192
  Volume of Distribution of HSG4112 (Vd/F)
Pharmacokinetic Assessment by Volume of Distribution of HSG4112 at Steady State | Hour 0 to 192
  Volume of Distribution of HSG4112 at Steady State (Vdss/F)
Safety and Tolerability Assessment by Adverse Event Monitoring | Day 1 to 9 following the last administration
  Number of participants with observed advese events
Safety and Tolerability Assessment by Number of Participants with Change in Vital Signs | Day 1 to 9 following the last administration
  Number of participants with clinically significant change in vital signs including blood pressure (mmHg) measured with blood pressure monitor, heart rate (beats per minute) measured with pulse oximeter, and body temperature (degrees Celcius) measured with thermometer
Safety and Tolerability Assessment by Number of Patients with Change in Physical Examination | Day 1 to 9 following the last administration
  Number of participants with clinically significant change in physical examination
Safety and Tolerability Assessment by Number of Participants with Change in Laboratory Test | Day 1 to 9 following the last administration
  Number of participants with clinically significant change in laboratory test assessed through hematology, blood biochemistry, urinalysis, and blood coagulation test
Safety and Tolerability Assessment by Number of Participants with Change in 12-Lead Electrocardiogram | Day 1 to 9 following the last administration
  Number of participants with clinically significant change in 12-lead electrocardiogram

SECONDARY OUTCOMES:
Pharmacodynamic Assessment by Change in Body Weight [Part 2] | Days 1 to 17, Day 18, Day 20, Day 22 post-dose before first meal
  Change in body weight
Pharmacodynamic Assessment by Change in Waist Circumference [Part 2] | Day 1, Day 8, Day 15, Day 22 post-dose before first meal
  Change in waist circumference
Pharmacodynamic Assessment by Change in Body Fat Mass [Part 2] | Day 1, Day 8, Day 15, Day 22 post-dose before first meal
  Change in body fat mass
Pharmacodynamic Assessment by Change in Body Fat Percentage [Part 2] | Day 1, Day 8, Day 15, Day 22 post-dose before first meal
  Change in body fat percentage
Pharmacodynamic Assessment by Change of Biomarkers [Part 2] | Day 1 and 14 pre-dose
  Measurement of biomarkers including leptin, adiponectin, insulin, C-peptide (connecting peptide), IL6 (interleukin 6), TNF-alpha (tumor necrosis factor alpha), and CCL2 (C-C motif ligand 2) from baseline to day of last dosing will be combined to assess the weight loss effect of HSG4112

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No